CLINICAL TRIAL: NCT01999023
Title: The Effects of Low Protein Formula on Renal Function, Oxidative Stress and Antioxidant Capacities in Patients With Chronic Kidney Disease
Brief Title: Effects of Low Protein Formula on Renal Function, Oxidative Stress and Antioxidant Capacities in CKD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SF13223
Record Dates: First submitted 2013-11-20; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational group (No Intervention): No intervention
- Dietary supplement (Experimental): Low protein formula formula (28.5 g) twice a day
  Interventions: Dietary Supplement: Low protein formula group

INTERVENTIONS:
Dietary Supplement: Low protein formula group — Low protein formula formula (28.5 g) twice a day
  Arms: Dietary supplement

SUMMARY:
Chronic renal disease is now the tenth leading cause of mortality Taiwan. It is worth to study the effect of low protein formula on the retardation of failing renal function, decrease plasma homocysteine and oxidative stress and further increase antioxidant capacities in patients with chronic kidney disease. The purpose of this study is going to investigate the effects of protein formula on renal function, homocysteine , oxidative stress and antioxidant capacities in patients with chronic kidney disease. One hundred and twenty patients with end stage renal disease (stage 2~4) who meet the inclusion criteria will be recruited from Taichung General Veterans Hospital, Taichung. Participant patients will be blinded and randomly assigned to either the placebo (n = 60) or low protein formula (n = 60) for 12 weeks. Data on demography, anthropometry and medical history will be collected, and fasting blood samples and 24 h urine samples will be obtained at week 0, 12 and 24 during intervention period. The levels of hematological, plasma and erythrocyte PLP, plasma pyridoxal and 4-pyridoxic acid, serum and erythrocyte folate, serum vitamin B-12, homocysteine, lipid peroxidation indicators, glutathione, total antioxidant capacity and antioxidant enzymatic will be measured. Twenty-four hour urine volume will be recorded and urine creatinine and urea nitrogen will be analyzed. Creatinine clearance rate will be measured. Hopefully, the results of this study could provide more pictures on beneficial effects of low protein formula on renal function, plasma homocysteine, oxidative stress and antioxidant capacities in patients with chronic kidney disease.

DETAILED DESCRIPTION:
Chronic renal disease is now the tenth leading cause of mortality Taiwan. It is worth to study the effect of low protein formula on the retardation of failing renal function, decrease plasma homocysteine and oxidative stress and further increase antioxidant capacities in patients with chronic kidney disease. The purpose of this study is going to investigate the effects of protein formula on renal function, homocysteine , oxidative stress and antioxidant capacities in patients with chronic kidney disease. This protocol is designed as a hospital-based blinded randomized placebo-controlled intervention trial. One hundred and twenty patients with end stage renal disease who meet the inclusion criteria will be recruited from Taichung General Veterans Hospital, Taichung. Participant patients will be blinded and randomly assigned to either the placebo (n = 60) or low protein formula (n = 60) for 12 weeks. Data on demography, anthropometry and medical history will be collected, and fasting blood samples and 24 h urine samples will be obtained at week 0, 12 and 24 during intervention period. The levels of hematological (red blood cell, hemoglobin, albumin, creatinine, urea nitrogen, total cholesterol, triglyceride, high and low density lipoprotein), plasma and erythrocyte PLP, plasma pyridoxal and 4-pyridoxic acid, serum and erythrocyte folate, serum vitamin B-12, homocysteine, lipid peroxidation indicators (serum malondialdehyde and oxidized low density lipoprotein), glutathione, total antioxidant capacity and antioxidant enzymatic activities (superoxide dismutase, glutathione peroxidase, glutathione S-transferase, glutathione reductase) will be measured. Twenty-four hour urine volume will be recorded and urine creatinine and urea nitrogen will be analyzed. Creatinine clearance rate will be measured. Hopefully, the results of this study could provide more pictures on beneficial effects of low protein formula on renal function, plasma homocysteine, oxidative stress and antioxidant capacities in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1) Diagnosed as stage 2 ~ 3 chronic kidney disease

Exclusion Criteria:

1. clinical unstable (i.e., systolic blood pressure < 90 mmHg, mean arterial blood pressure < 65 mmHg, fatal arrhythmia or the requirement of vasopressor to maintain blood pressure) or unconscious at any point during the study.
2. chronic diseases (i.e. liver disease, gastrointestinal diseases, alcoholism, cancer); or 3) being in pregnant or lactation.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Creatinine clearance rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan